CLINICAL TRIAL: NCT00641901
Title: A Study of Oral Health Care Education and Therapy to Reduce Gingivitis During Pregnancy
Brief Title: A Study to Evaluate Associations Between Gingivitis and Pregnancy Outcomes
Acronym: TRIUMPH
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Michael Reddy, DMD, Dean, School of Dentistry, University of Alabama at Birmingham
Other Study IDs: F070117004
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Pregnancy-associated Gingivitis
Keywords: gingivitis; pregnancy; pre-term birth
MeSH Terms: conditions — Gingivitis | interventions — Counseling; Lead; Toothbrushing; Diagnosis, Oral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples of venous blood and gingivial crevicular fluid (GCF)will be collected at baseline and at week-8.
  GCF samples will be harvested from two non-adjacent oral sites, flash-frozen in liquid nitrogen and stored at -70 degrees F. until batched testing. GCF samples will be analyzed for TNFalpha, IL1beta and IL 6 by Lumidex methodology.
  Blood samples will be analyzed for Serum Inflammatory markers, C-Reative Protein and inflammatory cytokines.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Pregnant women with gingivitis
  Interventions: Behavioral: counseling

INTERVENTIONS:
Behavioral: counseling — The 8-week study includes 3 visits to the dental facility at the Center for Women's Reproductive Health at UAB. Study visits are scheduled to coincide with pre-natal visits in the same facility.
  Each visit will include individually tailored one-to-one discussion with a dental professional coupled with a demonstration and instructions for using oral hygiene products. Home-care kits will be dispensed, to include a helpful digital video disk (DVD), a high-tech powered toothbrush, dental floss, toothpaste and alcohol-free mouth rinse and subjects will have their teeth professionally cleaned.
  First and final visits will include collection of gingival crevicular fluid and blood samples and subjects will complete pre and post study questionnaires.
  Other Names: Pre and Post-study questionnaires; Instructional DVD; Brushing and flossing instruction; Oral examination; Oral prophylaxis

SUMMARY:
Compelling evidence suggesting a possible link between maternal pregnancy-related periodontitis (gum disease) and spontaneous pre-term birth (PTB)makes effective management of oral health a relevant and significant obstetrical-dental issue.

The purpose of this pilot study is to determine whether intensive education and counseling can help pregnant women learn to maintain excellent oral health and in doing so reduce the severity of gingivitis and periodontitis during their pregnancy. Failure to effectively remove the plaque biofilm from the surface of teeth every day is the crucial event leading to the development of gingivitis and plaque-induced gingivitis is the most common form of periodontal disease in pregnant women.

We therefore hypothesize that patients can be taught to effectively modulate their own disease through intensive education and meticulous home care coupled with closely monitored behavior modification.

We believe this may be an effective approach toward improving oral health with the potential to reduce adverse pregnancy outcomes.

DETAILED DESCRIPTION:
Adverse pregnancy outcomes are significant personal and public health issues in the United States where approximately 12% of all births are pre-term (<37 weeks gestation). Care for these neonates accounts for over 5 million neonatal intensive care hospital stays each year and close to $6 Billion in annual health care costs. Premature delivery and low birth weight (LBW) are leading determinates of neonatal mortality and serious morbidity often leading to neurological and developmental restrictions in early childhood. Concomitant to these data are significant social and psychological consequences related to maternal and family distress and the effects of personal loss.

The role of maternal periodontitis as a potential stressor having detrimental effects on pregnancy outcomes is a relatively new area of investigation. Nevertheless, increasing evidence exists to support an association between maternal periodontal disease, a chronic anaerobic inflammatory condition of the oral cavity, and adverse pregnancy outcomes including pre-term birth (PTB) and fetal growth restriction. This is particularly true with very early-in-gestation delivery.

After adjusting for age, race, smoking and parity, a prospective study of over one-thousand pregnant women conducted at the University of Alabama at Birmingham (UAB) demonstrated that periodontal disease is associated with an increased risk of pre-term birth (PTB) by an odds ratio 4-7, depending on disease severity. These data showed a 55% prevalence of periodontal disease among this cohort; a much higher prevalence than had been reported in national surveys.

The mechanisms responsible for this association remain unclear. However, substantial data suggest that systemic inflammation, as measured by serum C-reactive protein and other inflammatory mediators may well underlie the observed associations.

Investigators hypothesize that links between maternal infections and pre-term bith involve microbes and host response to microbes that enter the uterine cavity during pregnancy. In cases of remote infection, such as periodontitis, this may occur via a blood-bourne route which triggers an alteration in the normal cytokine and hormone regulatory gestation that can result in premature labor, early rupture of membranes and preterm birth.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pregnancy between 16 and 24 weeks gestation
* Minimum of 20 natural teeth
* Gingival inflammation 50% of teeth

Exclusion Criteria:

* Multiple gestations
* Positive history for HIV infection, AIDS, Diabetes Mellitus
* Rampant untreated caries
* Concomitant Orthodontic treatment
* Medical condition that requires antibiotic prophylaxis prior to dental treatment
* Chronic use of medication that may cause gingival hypertrophy
* Chronic use of steroids
* Any obstetrical contraindication

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The Center for Women's Reproductive Heath at UAB
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2007-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Reduced gingival inflammation | 8 weeks

SECONDARY OUTCOMES:
Reduced pre-term birth | 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Reddy, DMD, DMSc, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The Center for Women's Reproductive Health at UAB, Birmingham, Alabama, United States

REFERENCES:
- [Background] Kramer MS. Determinants of low birth weight: methodological assessment and meta-analysis. Bull World Health Organ. 1987;65(5):663-737. PMID 3322602
- [Background] National Health Statistics. Health, United States, 1982 Washington DC:U S Government Printing Office; December 1982 DHHS publication (PHS) 83-1232
- [Background] Hamilton BE, Martin JA, Sutton PD; Centers for Disease Control and Prevention, National Center for Health Statistics. Births: preliminary data for 2003. Natl Vital Stat Rep. 2004 Nov 23;53(9):1-17. PMID 15622995
- [Background] Guyer B, Hoyert DL, Martin JA, Ventura SJ, MacDorman MF, Strobino DM. Annual summary of vital statistics--1998. Pediatrics. 1999 Dec;104(6):1229-46. doi: 10.1542/peds.104.6.1229. PMID 10585972
- [Background] Wienerroither H, Steiner H, Tomaselli J, Lobendanz M, Thun-Hohenstein L. Intrauterine blood flow and long-term intellectual, neurologic, and social development. Obstet Gynecol. 2001 Mar;97(3):449-53. doi: 10.1016/s0029-7844(00)01158-3. PMID 11239655
- [Background] Andrews WW, Hauth JC, Goldenberg RL. Infection and preterm birth. Am J Perinatol. 2000;17(7):357-65. doi: 10.1055/s-2000-13448. PMID 12141522
- [Background] Andrews WW, Goldenberg RL, Hauth JC. Preterm labor: emerging role of genital tract infections. Infect Agents Dis. 1995 Dec;4(4):196-211. PMID 8665085
- [Background] Goldenberg RL, Hauth JC, Andrews WW. Intrauterine infection and preterm delivery. N Engl J Med. 2000 May 18;342(20):1500-7. doi: 10.1056/NEJM200005183422007. No abstract available. PMID 10816189
- [Background] Hauth JC, Andrews WW, Goldenberg RL. Infection-related risk factors predictive of spontaneous birth. Prenat Neonat Med 1998;3:86-90
- [Background] Goepfert AR, Jeffcoat MK, Andrews WW, Faye-Petersen O, Cliver SP, Goldenberg RL, Hauth JC. Periodontal disease and upper genital tract inflammation in early spontaneous preterm birth. Obstet Gynecol. 2004 Oct;104(4):777-83. doi: 10.1097/01.AOG.0000139836.47777.6d. PMID 15458901
- [Background] Offenbacher S, Katz V, Fertik G, Collins J, Boyd D, Maynor G, McKaig R, Beck J. Periodontal infection as a possible risk factor for preterm low birth weight. J Periodontol. 1996 Oct;67(10 Suppl):1103-13. doi: 10.1902/jop.1996.67.10s.1103. PMID 8910829
- [Background] Jeffcoat MK, Geurs NC, Reddy MS, Cliver SP, Goldenberg RL, Hauth JC. Periodontal infection and preterm birth: results of a prospective study. J Am Dent Assoc. 2001 Jul;132(7):875-80. doi: 10.14219/jada.archive.2001.0299. PMID 11480640
- [Background] LOEE H. PERIODONTAL CHANGES IN PREGNANCY. J Periodontol (1930). 1965 May-Jun;36:209-17. No abstract available. PMID 14300227
- [Background] Arafat AH. Periodontal status during pregnancy. J Periodontol. 1974 Aug;45(8):641-3. doi: 10.1902/jop.1974.45.8.2.641. No abstract available. PMID 4529365
- [Background] Lopez NJ, Smith PC, Gutierrez J. Higher risk of preterm birth and low birth weight in women with periodontal disease. J Dent Res. 2002 Jan;81(1):58-63. doi: 10.1177/002203450208100113. PMID 11820369
- [Background] Lopez NJ, Smith PC, Gutierrez J. Periodontal therapy may reduce the risk of preterm low birth weight in women with periodontal disease: a randomized controlled trial. J Periodontol. 2002 Aug;73(8):911-24. doi: 10.1902/jop.2002.73.8.911. PMID 12211502
- [Background] Hill GB. Preterm birth: associations with genital and possibly oral microflora. Ann Periodontol. 1998 Jul;3(1):222-32. doi: 10.1902/annals.1998.3.1.222. PMID 9722706
- [Background] Gibbs RS. The relationship between infections and adverse pregnancy outcomes: an overview. Ann Periodontol. 2001 Dec;6(1):153-63. doi: 10.1902/annals.2001.6.1.153. PMID 11887458
- [Background] Romero BC, Chiquito CS, Elejalde LE, Bernardoni CB. Relationship between periodontal disease in pregnant women and the nutritional condition of their newborns. J Periodontol. 2002 Oct;73(10):1177-83. doi: 10.1902/jop.2002.73.10.1177. PMID 12416776
- [Background] Lopez NJ, Da Silva I, Ipinza J, Gutierrez J. Periodontal therapy reduces the rate of preterm low birth weight in women with pregnancy-associated gingivitis. J Periodontol. 2005 Nov;76(11 Suppl):2144-53. doi: 10.1902/jop.2005.76.11-S.2144. PMID 16277587
- [Background] Pepys MB, Hirschfield GM. C-reactive protein: a critical update. J Clin Invest. 2003 Jun;111(12):1805-12. doi: 10.1172/JCI18921. No abstract available. PMID 12813013
- [Background] Oppenheim J, Feldman M. Durham S, Hirano T, Vilcek J, Nicola N. Cytokine Reference: A Compendium of cytokines and other mediators of host defense. San Diego, CA Academic Press 2001 (vol 1)
- [Derived] Kaur M, Geisinger ML, Geurs NC, Griffin R, Vassilopoulos PJ, Vermeulen L, Haigh S, Reddy MS. Effect of intensive oral hygiene regimen during pregnancy on periodontal health, cytokine levels, and pregnancy outcomes: a pilot study. J Periodontol. 2014 Dec;85(12):1684-92. doi: 10.1902/jop.2014.140248. PMID 25079400